CLINICAL TRIAL: NCT05006911
Title: Pilocarpine, Brimonidine, Oxymetazoline Ophthalmic Compound Safety and Efficacy in Patients With Presbyopia
Brief Title: Pilocarpine, Brimonidine, Oxymetazoline (PBO) Compound to Control Presbyopia Symptoms
Acronym: PBO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Optall Vision (Other)
Responsible Party: Principal Investigator, Cesar Alejandro Sanchez Galeana, Principal Investigator, Optall Vision
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBOPC02
Record Dates: First submitted 2021-08-04; First posted 2021-08-16 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Pilocarpine; Brimonidine Tartrate; Oxymetazoline; Hyaluronic Acid; bromfenac

STUDY DESIGN:
Intervention Model Description: To determine safety and efficacy of a Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic Acid, Bromfenac compound to improve near uncorrected vision in healthy presbyopic patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PBOHB (Experimental): Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic Acid, Bromfenac to evaluate safety and efficacy to improve uncorrected near vision in healthy presbyopic patients
  Interventions: Drug: Pilocarpine, brimonidine, oxymetazoline, hyaluronic acid, bromfenac (PBOHB) compound

INTERVENTIONS:
Drug: Pilocarpine, brimonidine, oxymetazoline, hyaluronic acid, bromfenac (PBOHB) compound — To determine the safety and efficacy of a PBOHB compound in near vision of presbyopic patients.
  Other Names: PBOHB

SUMMARY:
Safety and Efficacy of Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac (PBOHB) ophthalmic compound to improve uncorrected near vision in healthy presbyopic patients one hour after instillation.

DETAILED DESCRIPTION:
To determine the safety and efficacy of a novel pharmacological compound of Pilocarpine, Brimonidine, Oxymetazoline, Hyaluronic acid, Bromfenac (PBOHB) to improve uncorrected near vision in healthy presbyopic patients one hour after binocular instillation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Presbyopic
* 40 - 60 years

Exclusion Criteria:

* Diabetics
* Previous eye surgery
* Previous eye disease
* > 0.50 myopia
* > 1.5 hyperopia or astigmatism

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Jaeger near uncorrected visual acuity improvement | 1 hour
  Measure uncorrected near vision change after binocular instillation of PBOHB compound

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Alejandro S Galeana, MD, Principal Investigator — Optall Vision
Locations (1):
- Optall Vision, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No